CLINICAL TRIAL: NCT00821912
Title: A Phase I/II Study on the Treatment With Taxotere in Combination With Xeloda in Patients With Metastatic Oesophageal Cancer or Cancer in the Cardia Region
Brief Title: TaxXel: Taxotere and Xeloda in Esophageal Cancer
Acronym: TaxXel
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Signe Friesland, MD, PhD, Karolinska University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TaxXel
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Cancer of the Esophagus; Gastric Cardia Carcinoma
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Docetaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Taxotere Xeloda (Experimental): Taxotere i.v. infusion on cycle day 1, 8 and 15 or cycle day 1 and 8 in an alternating 3 weekly schedule.
  Xeloda orally day 1-14 every 3 weeks.
  Interventions: Drug: Docetaxel; Drug: Capecitabine

INTERVENTIONS:
Drug: Docetaxel — 30 mg/m2, administered as a 30 min. i.v. infusion on cycle day 1, 8 and 15 or cycle day 1 and 8 in an alternating 3 weekly schedule
  Other Names: Taxotere
Drug: Capecitabine — 1650 mg/m2 /day orally b.i.d., day 1-14 every 3 weeks.
  Other Names: Xeloda

SUMMARY:
This is an open label, non-randomised, multicentre phase 1-2 study with a fixed dose of Taxotere in combination with Xeloda which is dose escalated during the first phase of the study (modified Fibonacci design) and fixed during the second phase.

The primary objective of the phase 1 part is to define the dose recommended for the Phase II part of the study. The primary objective is to determine the response rate.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma or adenocarcinoma of the oesophagus or cardia.
* Inoperable metastatic disease
* Performance status (WHO) of 0-2
* Measurable disease.
* Adequate hematological, liver and renal function.
* Signed informed consent.

Exclusion Criteria:

* CNS metastases
* Symptomatic peripheral neuropathy equal to or greater than NCI grade 2.
* Other concomitant serious illness or medical condition.
* Past or current history of malignant neoplasm other than oesophageal carcinoma.
* <18 years of age. Pregnant or lactating patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2006-03; Primary Completion 2012-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Response rate
  Response rate will be defined as the percentage of patients who achieve a complete response (CR) or partial response (PR).
  Duration of a CR or PR will be calculated from the time that measurement criteria are met for complete response or partial response until the first date that recurrent or progressive disease is objectively documented.

SECONDARY OUTCOMES:
CT scan | Every 9 weeks
Toxicity assessment | Every three weeks
Quality of life | Every three weeks

CONTACTS AND LOCATIONS:
Overall Officials: Signe Friesland, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (10):
- Norway (4):
  - Haukeland universitetssykehus, Bergen
  - Oslo universitetssykehus, Radiumhospitalet, Oslo
  - Oslo universitetssykehus, Ullevål, Oslo
  - St Olavs Hospital, Trondheim
- Sweden (6):
  - Linköping University Hospital, Linköping
  - Malmö General University Hospital, Malmo
  - Karolinska University Hospital, Dept of Oncology, Stockholm
  - Sundsvall County Hospital, Sundsvall
  - Uppsala Akademic Hospital, Uppsala
  - Västerås Central Hospital, Västerås